CLINICAL TRIAL: NCT00427830
Title: A Phase I Study of the Safety and Immunogenicity of a Recombinant MVA Vaccine Encoding a Secreted Antigen From M. Tuberculosis, Antigen 85A, Delivered Intradermally by a Needle Injection in Healthy Volunteers Who Have Previously Received BCG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB005
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2006-12

CONDITIONS: Tuberculosis
Keywords: Mycobacterium tuberculosis; 85A antigen; Recombinant Modified Vaccinia Ankara; Phase I study; Immunogenicity; BCG
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

INTERVENTIONS:
Biological: MVA85A

SUMMARY:
This is a phase I study to examine the safety and immunogenicity of MVA85A delivered intradermally into the deltoid region in volunteers who have recieved BCG in the past 20 years.

DETAILED DESCRIPTION:
This is a phase I study to examine the safety and immunogenicity of MVA85A delivered intradermally into the deltoid region in volunteers who have recieved BCG in the past 20 years

1. Selection of volunteers

Volunteers for the study will be recruited through advertisements. Each volunteer will have received an information sheet concerning the study and will have agreed to participate in writing. Volunteers will be given at least 48 hours between reading the information leaflet and agreeing to participate. Female volunteers will be told of the theoretical risk of congenital anomaly should they become pregnant during the study and only those who undertake to take precautions to avoid pregnancy during the study period will be eligible. Volunteers will give signed consent for their GP's to be notified about their participation in the trial. The GP will be faxed a letter on the day of screening and asked to reply if they know of a reason why the volunteer should not take part. The signed consent form will also be faxed with the letter.

2 Screening

Volunteers will be asked to sign the informed consent form for screening. The following will be performed:

* Medical history and examination
* Laboratory evaluations - including clinical chemistry, haematology, HLA typing, anti-vaccinia antibodies, anti-HBV antibodies, anti-HCV antibodies, anti-HIV antibodies
* Heaf test - to exclude prior exposure to TB
* Urinalysis and urine pregnancy test if female

  3 Inclusion Criteria
* Healthy adult aged 18-55 years.
* Normal medical history and physical examination.
* Normal urine dipstick, blood count, liver enzymes, and creatinine.

  4 Exclusion Criteria
  1. Exposure to TB at any point. Previous residence in a TB endemic area.
  2. Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness, psychiatric disorder, drug or alcohol abuse.
  3. Oral or systemic steroid medication or the use of immunosuppressive agents.
  4. Positive HIV antibody test, HCV antibody test or positive HBV serology except post-vaccination.
  5. Heaf test greater than Grade II
  6. Confirmed pregnancy
  7. Previous MVA immunisations

     5 Withdrawal Criteria

  <!-- -->

  1. Withdrawal of consent by subject for any reason
  2. Loss to follow-up
  3. Non-compliance with study procedures
  4. Protocol violation
  5. Serious adverse event (as defined in Appendix 3)
  6. Any other reason at discretion of the Principal Investigator
  7. Confirmed pregnancy during study period

     6 Immunisation

     On Day 0, subjects will receive a single intradermal injection of 5 x 107pfu in 0.1ml over the deltoid muscle. Subjects will be observed for an hour after all immunisations. Vital signs will be monitored at 30 and 60 minutes post-immunisation. Local reactions at the site of administration will be evaluated at 60 minutes.

     A photograph of the injection site may be taken at 48 hours (with written consent). The injection site will be reviewed 7 days after each immunization.

     Blood will be taken at the following time points: At the screening visit*, prior to the first vaccination, *1 week after the first vaccination, 2 weeks, 4 weeks, 8 weeks, *12 weeks, and 24 weeks after the vaccination. Up to 55 mls will be taken at any one time with the total being no more than 500 mls over the study period. *Samples taken on these dates will be tested for full blood count and biochemical screen. Immunological assays will be performed at all time points to determine vaccine immunogenicity. A pregnancy test will be performed prior to vaccination for female volunteers. Peripheral blood mononuclear cells will be prepared for cellular immunological assays to be performed without or following cryopreservation. Other serological measures of immune response, i.e. antibody titres, will be assayed on frozen plasma samples.

     All blood tests will be taken within 1-3 days of the due date as described in the schedule above.

     7 Endpoints

     The occurance and severity of local side-effects The occurance and severity of systemic side-effects The induction of T cell responses (as measured by an interferon-gamma Elispot assay).

     Proliferation assays and cytotoxic T cell assays will be performed on strong CD4+ and CD8+ responses respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-55 years.
* Normal medical history and physical examination.
* Normal urine dipstick, blood count, liver enzymes, and creatinine.

Exclusion Criteria:

* Exposure to TB at any point. Previous residence in a TB endemic area.
* Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness, psychiatric disorder, drug or alcohol abuse.
* Oral or systemic steroid medication or the use of immunosuppressive agents.
* Positive HIV antibody test, HCV antibody test or positive HBV serology except post-vaccination.
* Heaf test greater than Grade II
* Confirmed pregnancy
* Previous MVA immunisations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 2003-05; Study Completion 2005-01

PRIMARY OUTCOMES:
The occurance and severity of local and systemic side effects will be monitored. Vital signs and local reactions will be monitored at 30 and 60 minutes after each immunisation (and after 7 days).

SECONDARY OUTCOMES:
Immunogenicity will be measured: The induction of T cell responses (as measured by an interferon-gamma Elispot assay) will be performed on PBMCs from blood samples taken at the specified time points.
Proliferation assays and cytotoxic T cell assays will be performed on strong CD4+ and CD8+ responses respectively.
Antibody titres will be measured from frozen plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, MD and PhD, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Result] McShane H, Pathan AA, Sander CR, Keating SM, Gilbert SC, Huygen K, Fletcher HA, Hill AV. Recombinant modified vaccinia virus Ankara expressing antigen 85A boosts BCG-primed and naturally acquired antimycobacterial immunity in humans. Nat Med. 2004 Nov;10(11):1240-4. doi: 10.1038/nm1128. Epub 2004 Oct 24. PMID 15502839
- [Derived] Tanner R, Kakalacheva K, Miller E, Pathan AA, Chalk R, Sander CR, Scriba T, Tameris M, Hawkridge T, Mahomed H, Hussey G, Hanekom W, Checkley A, McShane H, Fletcher HA. Serum indoleamine 2,3-dioxygenase activity is associated with reduced immunogenicity following vaccination with MVA85A. BMC Infect Dis. 2014 Dec 3;14:660. doi: 10.1186/s12879-014-0660-7. PMID 25466778
- [Derived] Whelan KT, Pathan AA, Sander CR, Fletcher HA, Poulton I, Alder NC, Hill AV, McShane H. Safety and immunogenicity of boosting BCG vaccinated subjects with BCG: comparison with boosting with a new TB vaccine, MVA85A. PLoS One. 2009 Jun 16;4(6):e5934. doi: 10.1371/journal.pone.0005934. PMID 19529780
- [Derived] Pathan AA, Sander CR, Fletcher HA, Poulton I, Alder NC, Beveridge NE, Whelan KT, Hill AV, McShane H. Boosting BCG with recombinant modified vaccinia ankara expressing antigen 85A: different boosting intervals and implications for efficacy trials. PLoS One. 2007 Oct 24;2(10):e1052. doi: 10.1371/journal.pone.0001052. PMID 17957238